CLINICAL TRIAL: NCT00632827
Title: Treatment of Peripheral T-cell Lymphoma With Aggressive Induction Chemotherapy Followed by Autologous Stem Cell Transplant Using Denileukin Diftitox (Ontak) for In-vivo Purging and Post-Transplant Therapy: A Multicenter Phase II Clinical Trial
Brief Title: Treatment of PTCL With Aggressive Induction Therapy Followed by Autologous SCT Using Denileukin Diftitox (Ontak)
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Manufacturing shortage of both Diftitox and Doxil
Sponsor: University of California, San Francisco (Other)
Collaborators: Eisai Inc. (Industry); Washington University School of Medicine (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 072518; NCI-2011-01285 (Registry Identifier: NCI Clinical Trials Reporting Program (CTRP))
Record Dates: First submitted 2008-02-28; First posted 2008-03-11 (Estimated); Results first posted 2020-04-27 (Actual); Last update posted 2020-04-27 (Actual); Status verified 2020-04

CONDITIONS: Peripheral T-Cell Lymphoma
MeSH Terms: conditions — Lymphoma, T-Cell, Peripheral | interventions — Gemcitabine; Vinorelbine; liposomal doxorubicin; Granulocyte Colony-Stimulating Factor; pegfilgrastim; Cyclophosphamide; Vincristine; Leucovorin; Methotrexate; Doxorubicin; Cytarabine; Etoposide; etoposide phosphate; Carmustine; denileukin diftitox

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Treatment Plan (Experimental): (1) Induction Chemo A; Two 21-day cycles of Gemcitabine 1000 mg/m2 days (D) 1, 8, Navelbine 20 mg/m2 D1, D8; Doxil 15 mg/m2 Days 1 and 8, G-CSF Days 4-6 and 10-15 (2) Induction Chemo B: Two 21-day cycles of Cyclophosphamide 2000 mg/m2 day 1; Doxorubicin 50 mg/m2 day 1; Vincristine 1.4 mg/m2 day 1; Prednisone 100 mg/m2 days 1-5; Methotrexate 3000 mg/m2 IV over 4h day 15; Leucovorin rescue (3) Disease Evaluation (4) High-dose Consolidation Chemo, high dose Ara-C, Denileukin diftitox (Ontak) and Stem Cell Collection (5) Consolidation Cytarabine 2000 mg/m2 IV over 2 h q 12h days 1-4, Etoposide 40 mg/m2 continuous intravenous infusion (CIVI), days 1-4, Denileukin Diftitox (Ontak) 9 mcg/kg/day days 6-10, G-CSF 10 mcg/kg/day day 14+, Stem cell collection day 22 (6) Autologous Stem Cell Transplant Carmustine 550 mg/m2 day -6, Etoposide 60 mg/kg IV over 4h day -4, Cyclophosphamide 100 mg/kg day -2, Stem cell infusion D0 (7) Post-transplant: Denileukin Diftitox (Ontak) 18 mcg/kg/day days 1- 5
  Interventions: Drug: Gemcitabine; Drug: Navelbine; Drug: Doxorubicin Hydrochloride Liposome Injection; Drug: Granulocyte-colony stimulating factor (G-CSF); Drug: Pegfilgrastim; Drug: Cyclophosphamide; Drug: Vincristine; Drug: Leucovorin; Drug: Methotrexate; Drug: Doxorubicin Hydrochloride; Drug: Cytarabine; Drug: Etoposide; Drug: Carmustine; Drug: Denileukin diftitox

INTERVENTIONS:
Drug: Gemcitabine — Chemotherapy medication used to treat a number of types of cancer
  Other Names: Gemzar
Drug: Navelbine — Navelbine is an chemotherapy medication used to treat a number of types of cancer
  Other Names: Vinorelbine
Drug: Doxorubicin Hydrochloride Liposome Injection — Doxorubicin Hydrochloride Liposome Injection is an anti-cancer chemotherapy drug
  Other Names: Doxil
Drug: Granulocyte-colony stimulating factor (G-CSF) — G-CSF is a glycoprotein that stimulates the bone marrow to produce granulocytes and stem cells and release them into the bloodstream.
  Other Names: G-CSF
Drug: Pegfilgrastim — Colony-stimulating factor 3 (CSF 3) and, is a glycoprotein that stimulates the bone marrow to produce granulocytes and stem cells and release them into the bloodstream. May be used instead of G-CSF
  Other Names: Neulasta
Drug: Cyclophosphamide — Cancer medication that interferes with the growth and spread of cancer cells in the body
  Other Names: Cyclophosphamide 2000 MG; Cytoxan
Drug: Vincristine — Vincristine is a chemotherapy medication used to treat cancer. Vincristine works by stopping the cancer cells from separating into 2 new cells to stops the growth of the cancer
  Other Names: Vincrex; Vincasar PFS; Oncovin
Drug: Leucovorin — Leucovorin is used to prevent harmful effects of methotrexate when methotrexate is used to treat certain types of cancer.
  Other Names: Wellcovorin
Drug: Methotrexate — Methotrexate is a chemotherapy medication used to treat cancer
  Other Names: Rheumatrex; Trexall
Drug: Doxorubicin Hydrochloride — Doxorubicin Hydrochloride is a chemotherapy medication used to treat cancer
  Other Names: Adriamycin
Drug: Cytarabine — Medication used to treat acute myeloid leukemia (AML), acute lymphocytic leukemia (ALL), chronic myelogenous leukemia (CML), and non-Hodgkin's lymphoma
  Other Names: Ara-C; HiDAC
Drug: Etoposide — Etoposide is a is a chemotherapy medication used to treat cancer
  Other Names: Etopophos
Drug: Carmustine — Carmustine is a chemotherapy medication used to treat cancer
  Other Names: BCNU
Drug: Denileukin diftitox — Denileukin diftitox is an antineoplastic agent, an engineered protein combining Interleukin-2 and Diphtheria toxin. Denileukin diftitox could bind to Interleukin-2 receptors and introduce the diphtheria toxin into cells that express those receptors, killing the cells
  Other Names: Ontak

SUMMARY:
This study examines the use of denileukin diftitox (Ontak) for patients with peripheral T-cell lymphoma who are candidates for autologous stem cell transplants.

DETAILED DESCRIPTION:
This protocol proposes first to increase the proportion of patients who achieve adequate initial disease control and are able to proceed to autologous stem cell transplant (ASCT) in first complete or partial remission. It administers intensive and novel induction therapy.

Two cycles of gemcitabine, vinorelbine, Doxil (GND) will be used followed by two cycles of augmented dose Cyclophosphamide (CHOP) plus high-dose methotrexate (MTX). Patients will be restaged after two cycles of GND to assess response to GND alone and again after the second cycle of augmented CHOP/high-dose MTX.

Those achieving a remission status will receive intensive consolidation with HiDAC/etoposide followed by stem cell mobilization. A five-day course of denileukin diftitox (Ontak) will be administered at and will serve as an in vivo purge. This will be followed by autologous stem cell transplant.

Those not achieving partial remission or better following the four induction courses will receive 2 cycles of denileukin diftitox(Ontak) for 5 days. Those achieving partial remission or better to this regimen will go on to consolidation/mobilization and autologous stem cell transplant.

Post-transplant, denileukin diftitox will also be used as an additional module of therapy.

ELIGIBILITY:
Inclusion Criteria:

* Histologic diagnosis of any of the following:

  * Peripheral T-cell lymphoma not otherwise specified (PTCL-U),(IPI >2)
  * Angioimmunoblastic T-cell lymphoma (AILT) (IPI >2)
  * Non-primary cutaneous Alk-1-negative anaplastic large cell lymphoma
  * Extranodal natural killer (NK)/T lymphoma (Excluding stage I/II nasal disease)
  * Blastic NK cell lymphoma
  * Enteropathy type T-cell lymphoma
  * Cutaneous panniculitis-like T-cell lymphoma
  * Hepatosplenic T-cell lymphoma
* Measurable or assessable disease is not required.
* Age ≥ 18 and ≤ 70 years
* Previously untreated or 1 prior cycle of chemotherapy
* Creatinine < 2.0 mg/dL
* Total bilirubin < 2.0 mg/dL, aspartate aminotransferase (AST) < 3x upper limit of normal
* Patients who test positive for Hepatitis B surface Ag (HepBSAg) or Hepatitis C antibody (HepCAb) are eligible provided all of the following criteria are met:

  * bilirubin ≤ 2 x upper limit of normal;
  * aspartate aminotransferase (AST) ≤ 3 x upper limit of normal;
  * liver biopsy demonstrates ≤ grade 2 fibrosis and no cirrhosis.

Hepatitis B surface Ag(+) patients will be treated with lamivudine (3TC) or investigator's preferred antiviral regimen throughout protocol therapy and for 6-12 months thereafter.

* Neutrophils ≥ 1000/microlitre (uL) platelets > 100,000/uL
* HIV-negative
* Left ventricular ejection fraction (LVEF) of ≥ 45%
* No known hypersensitivity to denileukin diftitox or any of its components: diptheria toxin, interleukin-2, or excipients
* Non-pregnant, non-nursing: Treatment under this protocol would expose an unborn child to significant risks. Women and men of reproductive potential should agree to use an effective means of birth control.
* Patients with a "currently active" second malignancy, other than non-melanoma skin cancers are not eligible. (This includes Waldenstrom's Macroglobulinemia, since such patents have experienced transient increases inImmunoglobulin M (IgM) following initiation of rituximab, with the potential for hyperviscosity syndrome requiring plasmapheresis). Patients are not considered to have a "currently active" malignancy if they have completed anti-cancer therapy, and are considered by their physician to be at less than 30% risk of relapse.

Exclusion Criteria:

* PTCL-U / AILT with IPI 0 or 1 Extranodal NK/T nasal stage I/II T-lymphoblastic lymphoma Adult T-cell leukemia/lymphoma
* Adult T-cell leukemia/lymphoma

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 21 (Actual)
Dates: Start 2008-07-01 (Actual); Primary Completion 2014-06-23 (Actual); Study Completion 2016-06-23 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Lawrence Kaplan, MD, Principal Investigator — University of California, San Francisco
Locations (1):
- Washington University, St Louis, Missouri, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Groups:
- Treatment Plan: All patients will be given allopurinol 600 mg/day PO on day 1 of induction chemotherapy, and then 300 mg/day.
  Patients then receive two cycles of gemcitabine, vinorelbine, Doxil (GVD) followed by two cycles of augmented dose Cyclophosphamide (CHOP) plus high-dose Methotrexate (MTX). Patients were restaged after 2 cycles of GVD and again after the second cycle of augmented CHOP/high-dose MTX.
  Those achieving a remission status received intensive consolidation with Idarubicin/cytosine arabinoside(iDAC)/etoposide followed by stem cell mobilization and 5-day course of denileukin diftitox (Ontak) will be administered followed by autologous stem cell transplant.
  Those not achieving partial remission or better following the four induction courses will receive 2 cycles of denileukin diftitox(Ontak) for 5 days. Those achieving partial remission or better to this regimen moved to consolidation/mobilization and autologous stem cell transplant.
Period: Overall Study
Arm/Group | Treatment Plan
Started | 21
Received GVD | 21
Received M-CHOP | 18
Evaluated Post Stem Cell Transplant | 16
Completed | 11
Not Completed | 10
Not completed — Excluded after GVD (Not evaluable) | 2
Not completed — Death | 2
Not completed — Adverse Event | 5
Not completed — Lost to Follow-up | 1

BASELINE CHARACTERISTICS:
Groups:
- Treatment Plan: (1) Induction Chemo A; Two 21-day cycles of Gemcitabine 1000 mg/m2 days 1, 8, Navelbine 20 mg/m2 day 1, 8; Doxil 15 mg/m2 Days 1, 8, Granulocyte-colony stimulating factor(G-CSF) Days 4-6 and 10-15 (2) Induction Chemo B: Two 21-day cycles of Cyclophosphamide 2000 mg/m2 day 1; Doxorubicin 50 mg/m2 day 1; Vincristine 1.4 mg/m2 day 1; Prednisone 100 mg/m2 days 1-5; Methotrexate 3000 mg/m2 IV over 4h day 15; Leucovorin rescue (3) Disease Evaluation (4) High-dose Consolidation Chemo, high dose Ara-C, Denileukin diftitox (Ontak) and Stem Cell Collection (5) Consolidation Cytarabine 2000 mg/m2 IV over 2 h q 12h days 1-4, Etoposide 40 mg/m2 continuous intravenous infusion days 1-4, Denileukin Diftitox (Ontak) 9 mcg/kg/day days 6-10, G-CSF 10 mcg/kg/day day 14+, Stem cell collection day 22 (6) Autologous Stem Cell Transplant Carmustine 550 mg/m2 day 1-6, Etoposide 60 mg/kg IV over 4h day -4, Cyclophosphamide 100 mg/kg day -2, Stem cell infusion day 0 (7) Post-transplant: Denileukin diftitox
Arm/Group | Treatment Plan
Number analyzed (Participants) | 21
Age, Continuous [Median (Full Range); unit: years] | 58 [26 to 68]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 8
  Male | 13
Region of Enrollment [Number; unit: participants]
  United States | 21
Histology [Count of Participants; unit: Participants]
  Angioimmunoblastic T-cell lymphoma (AILT) | 8
  Peripheral T-cell lymphoma (PTCL) not classified | 9
  Enteropathy-associated T-cell lymphoma | 1
  Subcutaneous panniculitis-like T-cell Lymphoma | 1
  Hepato-Splenic gamma-delta T-cell Lymphoma | 1
  Anaplastic large cell lymphoma, ALK- | 1
Extranodal Sites [Count of Participants; unit: Participants]
  Bone Marrow | 7
  Skin | 3
  Bone | 3
  Gastrointestinal | 2
  Lung | 1
  Liver | 1
  Thyroid | 1
  No extranodal site | 3
Disease Stage [Count of Participants; unit: Participants] — The American Joint Committee on Cancer (AJCC) and the International Union for Cancer Control (UICC) maintain the classification system as a tool for doctors to stage different types of cancer based on certain standards. The stage refers to the extent of your cancer, such as how large the tumor is, and if it has spread. A cancer is always referred to by the stage it was given at diagnosis and is assigned a roman numeral from 0 to IV, where stage 0 is the least severe and stage 4 (IV) is the more severe and the cancer is more advanced than in the lower stages
  Participants
    Stage I/II | 0
    Stage III | 7
    Stage IV | 14
Lactate Dehydrogenase (LDH)> normal [Count of Participants; unit: Participants] | 19
International prognostic index (IPI) score [Count of Participants; unit: Participants] — The International Prognostic Index (IPI) is a clinical tool developed by oncologists to aid in predicting the prognosis of patients. The score range is 0-5 with lower scores indicating a lower risk of death and higher scores indicating a greater risk of death.
  Participants
    Score of 2 | 6
    Score of 3 | 12
    Score of >=4 | 3

OUTCOME MEASURES:

1. Primary Outcome: Progression Free Survival
Description: Progression-Free Survival will be defined the percentage of participants alive and progression-free at median follow up of 25 months. Patients will be routinely followed for disease progression and those who die without a reported prior progression will be considered to have progressed on the day of their death. Patients who did not progress or die will be censored at the day of their last treatment assessment. Patients who have not received study regimen or did not have on-study treatment assessments will be censored on the day they entered the trial. Patients who receive chemotherapy for reasons other than documented progression of disease or clinical progression without documented progression will be censored on the earliest date of subsequent therapy
Time Frame: Up to 3 years
Measure: Number; unit: percentage of partcipants
Groups:
- Treatment Plan: (1) Induction Chemo A; Two 21-day cycles of Gemcitabine 1000 mg/m2 days 1, 8, Navelbine 20 mg/m2 day 1, 8; Doxil 15 mg/m2 Days 1 and 8, G-CSF Days 4-6 and 10-15 (2) Induction Chemo B: Two 21-day cycles of Cyclophosphamide 2000 mg/m2 day 1; Doxorubicin 50 mg/m2 day 1; Vincristine 1.4 mg/m2 day 1; Prednisone 100 mg/m2 days 1-5; Methotrexate 3000 mg/m2 IV over 4h day 15; Leucovorin rescue (3) Disease Evaluation (4) High-dose Consolidation Chemo, high dose Ara-C, Denileukin diftitox (Ontak) and Stem Cell Collection (5) Consolidation Cytarabine 2000 mg/m2 IV over 2 h q 12h days 1-4, Etoposide 40 mg/m2 continuous intravenous infusion days 1-4, Denileukin Diftitox (Ontak) 9 mcg/kg/day days 6-10, G-CSF 10 mcg/kg/day day 14+, Stem cell collection day 22 (6) Autologous Stem Cell Transplant Carmustine 550 mg/m2 day -6, Etoposide 60 mg/kg IV over 4h day -4, Cyclophosphamide 100 mg/kg day -2, Stem cell infusion day 0 (7) Post-transplant: Denileukin Diftitox (Ontak) 18 mcg/kg/day days 1- 5
Arm/Group | Treatment Plan
Number analyzed (Participants) | 21
percentage of partcipants | 65

2. Secondary Outcome: Overall Survival Rate
Description: Overall Survival will be defined the percentage of participants alive at median follow up of 25 months. If the patient is lost to follow-up, survival will be censored on the last date the patient was known to be alive. The analysis is expected to occur up to 60 months after the first patient is entered the trial.
Time Frame: Up to 5 years
Measure: Number; unit: percentage of participants
Arm/Group | Treatment Plan
Number analyzed (Participants) | 21
percentage of participants | 75

3. Secondary Outcome: Complete Response Rate
Description: The complete response rate will be defined as the total number of patients who have defined complete response using study regimen (intensive induction therapy/progressive chemotherapy/stem cell rescue), divided by the number of patients entered in the trial using response-evaluable patients.
Time Frame: Up to 3 years
Measure: Count of Participants; unit: Participants
Groups:
- Treatment Plan: All patients will be given allopurinol 600 mg/day PO on day 1 of induction chemotherapy, and then 300 mg/day.
  Patients then receive two cycles of gemcitabine, vinorelbine, Doxil (GND) followed by two cycles of augmented dose Cyclophosphamide (CHOP) plus high-dose Methotrexate (MTX). Patients were restaged after 2 cycles of GND and again after the second cycle of augmented CHOP/high-dose MTX.
  Those achieving a remission status received intensive consolidation with iDAC/etoposide followed by stem cell mobilization and 5-day course of denileukin diftitox (Ontak) will be administered followed by autologous stem cell transplant.
  Those not achieving partial remission or better following the four induction courses will receive 2 cycles of denileukin diftitox(Ontak) for 5 days. Those achieving partial remission or better to this regimen moved to consolidation/mobilization and autologous stem cell transplant.
Arm/Group | Treatment Plan
Number analyzed (Participants) | 21
Participants | 14

4. Secondary Outcome: Median Time to Response
Description: The time to response is measured from the time measurement criteria are met for complete response or partial response (whichever is first recorded) until the first date that recurrent or progressive disease is objectively documented (taking as reference for progressive disease the smallest measurements recorded since the treatment started) in months.
Time Frame: Up to 2 years
Measure: Median (Full Range); unit: months
Arm/Group | Treatment Plan
Number analyzed (Participants) | 21
months | 3.0 [1.4 to 19.4]

ADVERSE EVENTS:
Time Frame: Up to 5 years
Arm/Group | Treatment Plan
All-Cause Mortality (participants affected / at risk) | 7/21
Serious Adverse Events (participants affected / at risk) | 21/21
Other Adverse Events (participants affected / at risk) | 11/21
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Treatment Plan (N=21)
Cytopenia (Blood and lymphatic system disorders) | 21 (21)
Febrile neutropenia (Blood and lymphatic system disorders) | 11 (11)
Sepsis/Bacteremia (Infections and infestations) | 6 (6)
Capillary leak syndrome (Vascular disorders) | 1 (1)
Renal Failure (Renal and urinary disorders) | 1 (1)
Hypotension (Cardiac disorders) | 4 (4)
Cholecystitis (Hepatobiliary disorders) | 1 (1)
Infection with normal ANC or Grade 1 or 2 neutrophils (Infections and infestations) | 3 (3)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Treatment Plan (N=21)
Diarrhea (Gastrointestinal disorders) | 2 (4)
Pneumonitis/pulmonary infiltrates (Respiratory, thoracic and mediastinal disorders) | 2 (2)
Liver Function abnormalities (Metabolism and nutrition disorders) | 7 (7)

LIMITATIONS AND CAVEATS:
Enrollment was terminated prematurely due to manufacturing shortages of Doxil and Denileukin Diftitox (Ontak). All eligible patients who received at least one dose of study regimen were included in the analyses

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No